CLINICAL TRIAL: NCT00068120
Title: ORWH:SCOR - Sex/Gender Factors Affecting Women's Health
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: ORWHSCOR-dk64540 (compltd)
Record Dates: First submitted 2003-09-08; First posted 2003-09-09 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Urinary Tract Infection
Keywords: Urinary tract infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This project is the clinical project of a Specialized Center of Research (SCOR) proposal which is designed to further our understanding of urinary tract infection (UTI) in women. Acute uncomplicated urinary tract infections (UTIs) occur in an estimated 7-11 million women each year, and the annual costs of caring for these women are thought to approach $1.6 billion. Approximately 20-30% of women suffer from frequent recurrent infections. UTIs in young women result in substantial symptoms, time lost from work, and medical costs. An improved understanding of the mechanisms underlying UTIs could result in new approaches to their prevention and reduced numbers of women with infections and the amount of antibiotics use.

In this project we seek a better understanding of the causes of UTI. Most experts believe that vaginal colonization with UTI-causing bacteria from the rectal flora precedes colonization of the urethra (the tube from the bladder for urination) and bladder and subsequent UTI, but the relationships between these events has not been established. Moreover, recent information from studies in mice strongly suggest that persistent bladder infection follows an initial bladder infection.

In this project, we will prospectively follow a large group of women with recurrent UTI to determine: 1) the relationships in time between vaginal colonization with a UTI-causing bacteriuria, asymptomatic bacteriuria (bacteria in the bladder but without any UTI symptoms) and symptomatic UTI, and 2) the presence of persistent bacteria in the bladder following the symptomatic UTI at entry into the study and whether such bacteria are related to later UTIs that are caused by the same bacteria that caused the UTI at entry into the study. We will thus be able to determine the relative importance of vaginal colonization vs. persistent infection of the bladder as the origin of the bacteria causing recurrent UTI.

UTI-causing bacteria cultured from women with symptomatic UTI and asymptomatic bacteriuria will undergo studies by Dr. Scott Hultgren's group at Washington University in Project 1 to identify unique genes that may help us understand why some bacteria cause symptoms and others do not. The effect of bacteria causing UTI in these women on host response will also be determined by studies by Dr. Jeff Gordon's laboratory at Washington University in Project 3.

A better understanding of the molecular and epidemiologic basis of UTI is critical in developing the best possible prevention and management strategies.

ELIGIBILITY:
* Healthy women with bladder infection who have a history of at least one previous UTI in the past 12 months.
* Women must be able to provide written informed consent.
* They must not be pregnant or planning on becoming pregnant in the next 3 months, have no chronic illness, have no known anatomic or functional abnormalities of the urinary tract and not have any symptoms suggestive of kidney infection.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Hall Health Primary Care Center, Seattle, Washington, United States